CLINICAL TRIAL: NCT01048411
Title: Multicenter Randomized Controlled Trial to Investigate the Influence of the Homeopathic Remedy 'Naja-comp' on Stroke Therapy in Geriatric Rehabilitation
Brief Title: Trial to Investigate the Influence of the Homeopathic Remedy Naja-comp on Stroke Therapy in Geriatric Rehabilitation
Acronym: naja-comp
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Erlangen-Nürnberg Medical School (Other)
Responsible Party: Prof. Dr. Cornel Sieber, University of Erlangen-Nuernberg, Institute for Biomedicine of Aging
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: naja-comp-1-trial; 2004-001760-46 (EudraCT Number)
Record Dates: First submitted 2009-10-07; First posted 2010-01-13 (Estimated); Last update posted 2020-12-14 (Actual); Status verified 2020-12

CONDITIONS: Stroke
Keywords: stroke rehabilitation; outcome; barthel-index; geriatrics; elderly
MeSH Terms: conditions — Stroke | interventions — Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Naja-comp. (Active Comparator): s.c. injection of naja comp (homeopathic remedy) three times a week
  Interventions: Drug: Naja-comp.
- Placebo (Placebo Comparator): s.c. injection of placebo (NaCl-solution) three times a week
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Naja-comp. — homeopathic remedy
  Other Names: Naja compositum
  Arms: Naja-comp.
Drug: Placebo — s.c. injection of NaCl-solution three times a week
  Other Names: NaCl 0.9%
  Arms: Placebo

SUMMARY:
The homeopathic remedy 'naja-comp' will improve functional outcome measured by the Barthel-Index.

The homeopathic remedy 'naja-comp' will decrease complications during geriatric rehabilitation measured by rate of unplanned discharge to hospital.

DETAILED DESCRIPTION:
Secondary outcome for functional improvement are Scandinavian Stroke Scale, 4D+S-Scale and Timed-Up&Go-Test.

ELIGIBILITY:
Inclusion Criteria:

* stroke within 60 days after onset

Exclusion Criteria:

* stroke by injury or tumor
* stroke older than 60 days
* missing consent for participation
* participation at other clinical trials

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 344 (Actual)
Dates: Start 2006-01; Primary Completion 2009-08 (Actual); Study Completion 2009-08 (Actual)

PRIMARY OUTCOMES:
barthel-index | baseline, 21st day of rehabilitation
rate of unplanned discharge to hospital care | until day 21 of rehabilitation

SECONDARY OUTCOMES:
Scandinavian Stroke Scale, 4D+S-Scale, Timed-Up&Go-Test | baseline, 21st day of rehabilitation

CONTACTS AND LOCATIONS:
Overall Officials: Cornel Sieber, Professor, Study Chair — Univerity of Erlangen-Nuernberg, Director of the Institute for Biomedicine of Aging
Locations (3):
- Germany (3):
  - KWA Stift Rottal, Bad Griesbach, Bavaria
  - Alexander von Humdoldt-Klijnik, Bad Steben, Bavaria
  - Kreiskrankenhaus Haag - Fachklinik für Geriatrische Rehabilitation, Haag in Oberbayern, Bavaria